CLINICAL TRIAL: NCT01986088
Title: A Multicentre, Double Blind, Double Dummy, Parallel Group, Placebo Controlled, Study of Two Dose Levels of Oral Eletriptan and Two Dose Levels Oral Sumatriptan Given for the Acute Treatment of Migraine(With and Without Aura).
Brief Title: Eletriptan vs Sumatriptan: A Double-blind, Placebo-controlled, Multiple Migraine Attack Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A160-318
Record Dates: First submitted 2013-11-11; First posted 2013-11-18 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Migraine With or Without Aura
MeSH Terms: interventions — eletriptan; Sumatriptan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Eletriptan 40 mg (Experimental)
  Interventions: Drug: Eletriptan 40 mg
- Eletriptan 80 mg (Experimental)
  Interventions: Drug: Eletriptan 80 mg
- Sumatriptan 50 mg (Experimental)
  Interventions: Drug: Sumatriptan 50 mg
- Sumatriptan 100 mg (Experimental)
  Interventions: Drug: Sumatriptan 100 mg

INTERVENTIONS:
Drug: Placebo — matching placebo
  Arms: Placebo
Drug: Eletriptan 40 mg — 40mg oral
  Arms: Eletriptan 40 mg
Drug: Eletriptan 80 mg — 80mg oral
  Arms: Eletriptan 80 mg
Drug: Sumatriptan 50 mg — 50mg oral
  Arms: Sumatriptan 50 mg
Drug: Sumatriptan 100 mg — 100mg oral
  Arms: Sumatriptan 100 mg

SUMMARY:
A previously published, placebo-controlled, head-to-head comparator study found eletriptan to have superior efficacy to oral sumatriptan 100 mg in treating a single acute migraine attack. The goal of the current study was to extend the findings of that study by examining the efficacy of eletriptan compared with both 50- and 100-mg doses of sumatriptan; and to evaluate the comparative efficacy of eletriptan and sumatriptan across additional important clinical outcomes. In particular, early response (at 1 hour), sustained response (without need for additional treatment) at 24 hours, and consistency of response across multiple attacks were examined.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients were men and women with a minimum age limit of 18 years of age (in Canada there was also an age limit of 65 years) who were expected to have at least one attack of migraine with or without aura, as defined by the International Headache Society (IHS) criteria,15 every 6 weeks.
* Patients had to be capable of taking study medication as outpatients and recording the effects.

Exclusion Criteria:

* Pregnant or breast-feeding women and those not using adequate contraception were excluded from the trial.
* Patients with frequent nonmigrainous headache, atypical migraine that had not previously responded to therapy, migraine with prolonged aura, familial hemiplegic migraine, basilar migraine, or migrainous infarction were excluded from the trial.

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1008 (Actual)
Dates: Start 1996-11; Primary Completion 1998-01 (Actual); Study Completion 1998-01 (Actual)

PRIMARY OUTCOMES:
Headache response at 1 hour after treatment of the first attack. | 1 hour
  Headache response was defined as improvement from a severe or moderate headache at baseline to either a mild or absent headache post-dose.

SECONDARY OUTCOMES:
Headache severity | .5, 1, 2, 4 and 24 hours
Pain-free response | .5, 1, 2, 4 and 24 hours
Functional response | .5, 1, 2, 4 and 24 hours
Presence or absence of nausea, photophobia, and phonophobia | .5, 1, 2, 4 and 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A160-318&StudyName=Eletriptan%20vs%20Sumatriptan%3A%20A%20double-blind%2C%20placebo-controlled%2C%20multiple%20migraine%20attack%20study